CLINICAL TRIAL: NCT03449199
Title: A Randomized, Placebo-Controlled, Double-Blind, Multicenter, Phase 2 Study to Assess Safety, Tolerability, and Renal Effects of TMX-049 in Subjects With Type 2 Diabetes and Albuminuria
Brief Title: Phase 2 Study of TMX-049 in Subjects With Type 2 Diabetes and Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teijin America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-049DN-201
Record Dates: First submitted 2018-02-09; First posted 2018-02-28 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; XO inhibitor; UACR
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TMX-049 40 mg QD (Once Daily) (Experimental): TMX-049: 40 mg of TMX-049 to be taken orally, once daily
  Interventions: Drug: TMX-049
- TMX-049 200 mg QD (Once Daily) (Experimental): TMX-049: 200 mg of TMX-049 to be taken orally, once daily
  Interventions: Drug: TMX-049
- TMX-049 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TMX-049 — A certain dose of TMX-049 to be taken orally, once daily
  Arms: TMX-049 200 mg QD (Once Daily); TMX-049 40 mg QD (Once Daily)
Drug: Placebo — Matching placebo to be taken orally, once daily
  Arms: TMX-049 Placebo

SUMMARY:
The primary objective of this study is to assess the effect of 2 dose levels of TMX-049 on urinary albumin excretion in subjects with Type 2 diabetes and albuminuria (a urinary albumin-to-creatinine ratio (UACR) 200 to 3000 mg/g and an estimated glomerular filtration rate (eGFR) ≥30 ml/min/1.73m2). Effects of each TMX-049 dose on UACR will be assessed in terms of ratios using log-transformed UACR at Baseline and after a 12-week period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes treated with ≥1 glucose-lowering medication for at least 12 months
* UACR 200 to 3000 mg/g
* eGFR ≥30 ml/min/1.73m2
* Treated with at least the minimal recommended dose of an angiotensin converting enzyme inhibitor (ACEI) or an angiotensin II receptor blocker (ARB), but not both

Exclusion Criteria:

* History of Type 1 diabetes
* Women who are breast feeding
* Treatment with any uric acid-lowering therapy within previous 2 weeks
* History of intolerance to any XO (xanthine oxidase) inhibitor
* History of a gout flare requiring pharmacologic treatment
* History or presence of tophaceous gout
* History of immunosuppressant treatment for any known or suspected renal disorder
* History of a non-diabetic form of renal disease
* Glycosylated hemoglobin (HbA1c) >11%
* sUA <4.0 mg/dL or >10.0 mg/dL
* Positive urinary pregnancy test
* Dialysis for acute renal failure within previous 6 months
* Renal allograft in place or a scheduled kidney transplant within the next 22 weeks
* Congenital or acquired solitary kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cressman, D.O., Study Director — Covance
Locations (55):
- United States (55):
  - AKDHC Medical Research Services, LLC, Flagstaff, Arizona
  - Aventiv Research Inc., Mesa, Arizona
  - Comprehensive Research Institute, Alhambra, California
  - California Kidney Specialists, Covina, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Diabetes Associates Medical Group, Orange, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - California Kidney Specialists, San Dimas, California
  - North America Research Institute, San Dimas, California
  - Leon Medical Research, Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Endocrine Associates of Florida, P.A., Ocoee, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Nephrology Associates, PC, Augusta, Georgia
  - Southeastern Clinical Research Institute, Augusta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Llc, Meridian, Idaho
  - Associate in Endocrinology, Elgin, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Community Hospital of Anderson and Madison County, Inc., Anderson, Indiana
  - Iowa Kidney Physicians, Des Moines, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - My Kidney Center, LLC., Manhattan, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Four Rivers Clincial Research, Paducah, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Baton Rouge, Louisiana
  - Biolab Research LLC, Rockville, Maryland
  - Aa Mrc Llc, Flint, Michigan
  - Elite Research Center LLC, Flint, Michigan
  - Endocrine Consultants of Mid Michigan, Flint, Michigan
  - Seacost Kidney & Hypertension Specialists, Portsmouth, New Hampshire
  - Albany Medical College, Division of Community Endocinology, Albany, New York
  - Randolph Health Internal Medicine, Asheboro, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc. Centennial Health, PC, Oklahoma City, Oklahoma
  - Detweiler Family Medicine & Associates, PC, Lansdale, Pennsylvania
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Texas Health Physicians Group, Dallas, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - Rockwood Medical Clinic, Fort Worth, Texas
  - Endocrine Associates, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - The Endocrine Center, Houston, Texas
  - Pioneer Research Solutions INC, Houston, Texas
  - Houston Nephrology Research, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - BFHC Research, San Antonio, Texas
  - Carl R. Meisner Medical Clinic, PLLC, Sugar Land, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia

REFERENCES:
- [Derived] Bakris GL, Mikami H, Hirata M, Nakajima A, Cressman MD. A Non-purine Xanthine Oxidoreductase Inhibitor Reduces Albuminuria in Patients with DKD: A Randomized Controlled Trial. Kidney360. 2021 Jun 30;2(8):1240-1250. doi: 10.34067/KID.0001672021. eCollection 2021 Aug 26. PMID 35369650

RESULTS

PARTICIPANT FLOW:
Groups:
- TMX-049 40mg QD: TMX-049: 40mg of TMX-049 to be taken orally, once daily
- TMX-049 200mg QD: TMX-049: 200 mg of TMX-049 to be taken orally, once daily
Period: Overall Study
Arm/Group | TMX-049 Placebo | TMX-049 40mg QD | TMX-049 200mg QD
Started | 42 | 44 | 44
Completed | 41 | 43 | 42
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TMX-049 40 mg QD: TMX-049: 40 mg of TMX-049 to be taken orally, once daily
- TMX-049 200 mg QD: TMX-049: 200 mg of TMX-049 to be taken orally, once daily
- Total: Total of all reporting groups
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD | Total
Number analyzed (Participants) | 42 | 43 | 44 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10.3) | 66 (10.7) | 68 (10) | 66 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 18 | 53
  Male | 24 | 26 | 26 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 8 | 15
  White | 32 | 38 | 35 | 105
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 90.1 (19.81) | 95.9 (20.58) | 98.8 (23.63) | 95.0 (21.57)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (6.00) | 33.6 (6.57) | 34.3 (7.26) | 32.2 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Log-transformed Urinary Albumin-to-creatinine Ratio (UACR) at Week 12
Description: UACR from Baseline to Weeks 2, 6, 12, and 16(Follow-up) were measured. The change from baseline at Week 12 in log-transformed UACR was analyzed and reported as a primary outcome.
Time Frame: Baseline and Week 12
Population: Modified Intention-to-Treat (mITT) Population consisted of all randomized subjects who had at least 1 post-randomization UACR assessment. Subjects in the mITT Population were analyzed according to their randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: Log(mg/g)
Groups:
- TMX-049 Placebo: Placebo: Matching placebo to be taken orally, once daily, for 12 weeks
- TMX-049 40 mg QD: TMX-049: 40 mg of TMX-049 to be taken orally, once daily for 12 weeks
- TMX-049 200 mg QD: TMX-049: 200 mg of TMX-049 to be taken orally, once daily for 12 weeks
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 43 | 44
Log(mg/g) | -0.10 (0.153) | -0.15 (0.151) | -0.53 (0.150)
Statistical Analysis 1: Comparison: TMX-049 Placebo vs TMX-049 40 mg QD; Change from baseline in log-transformed UACR was analyzed using an ANCOVA model with randomized treatment, and randomization strata of sUA and UACR as independent variables. The last observation carried forward imputation was used for missing data. In this study, multiplicity was not considered since the study objective is exploratory; Test type: Superiority; p = 0.7953, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.44 to 0.34]
Statistical Analysis 2: Comparison: TMX-049 Placebo vs TMX-049 200 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0311, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.82 to -0.04]

2. Secondary Outcome: Changes in Estimated Glomerular Filtration Rate (GFR)
Description: Estimated Glomerular Filtration Rate from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured. The eGFR (estimated glomerular filtration rate) was calculated using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula based on the serum creatinine measurement.
Time Frame: Baseline and Week 2, 6, 12, 16 (Follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ml/min/1.73 m^2
Groups:
- TMX-049 Placebo: Placebo: Matching placebo to be taken orally, once daily for 12 weeks
- TMX-049 40 mg QD: TMX-049:40 mg of TMX-049 to be taken orally, once daily for 12 weeks
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 43 | 44
ml/min/1.73 m^2
  Visit 4 (Week 2): number analyzed (Participants) | 42 | 42 | 44
  Visit 4 (Week 2) | -0.02 (1.591) | 0.98 (1.601) | 0.18 (1.561)
  Visit 5 (Week 6) | -1.41 (1.757) | -1.06 (1.732) | 0.00 (1.724)
  Visit 6/ET (Week 12) | -2.34 (1.585) | -0.62 (1.563) | 1.09 (1.556)
  Visit 7/Follow up (Week 16) | -2.39 (1.726) | 1.57 (1.702) | 0.99 (1.695)
Statistical Analysis 1: Comparison: TMX-049 Placebo vs TMX-049 40 mg QD; For Week 12 (visit of the primary outcome), ANCOVA model with treatment, randomization strata of sUA and UACR levels as independent variables, Baseline eGFR as covariate is fitted. The last observation carried forward imputation was used for missing data; Test type: Superiority; p = 0.4055, ANCOVA; LS Mean Difference = 1.71, 95% CI 2-sided [-2.35 to 5.78]
Statistical Analysis 2: Comparison: TMX-049 Placebo vs TMX-049 200 mg QD; For Week 12 (visit of the primary outcome), an ANCOVA model with treatment, randomization strata of sUA and UACR levels as independent variables, Baseline eGFR as covariate is fitted. The last observation carried forward imputation was used for missing data; Test type: Superiority; p = 0.0960, ANCOVA; LS Mean Difference = 3.42, 95% CI 2-sided [-0.62 to 7.46]

3. Secondary Outcome: Changes in Serum Uric Acid (sUA)
Description: Serum Uric Acid from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured in order to explore the sUA (Serum Uric Acid) lowering effect in DKD (diabetic kidney disease) patients and the relationship between sUA and efficacy to DKD.
Time Frame: Baseline and Week 2, 6, 12, 16 (Follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 43 | 44
mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 42 | 42 | 44
  Visit 4 (Week 2) | -0.03 (0.238) | -2.57 (0.240) | -3.54 (0.234)
  Visit 5 (Week 6) | -0.22 (0.256) | -2.54 (0.252) | -3.34 (0.251)
  Visit 6/ET (Week 12) | -0.07 (0.269) | -2.51 (0.266) | -3.30 (0.265)
  Visit 7/Follow up (Week 16) | 0.21 (0.190) | -0.13 (0.188) | -0.33 (0.187)
Statistical Analysis 1: Comparison: TMX-049 Placebo vs TMX-049 40 mg QD; For Week 12 (visit of the primary outcome), an ANCOVA model with treatment, randomization strata of UACR levels as independent variables is fitted. The last observation carried forward imputation was used for missing data; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.43, 95% CI 2-sided [-3.13 to -1.74]
Statistical Analysis 2: Comparison: TMX-049 Placebo vs TMX-049 200 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -3.23, 95% CI 2-sided [-3.91 to -2.54]

4. Secondary Outcome: Changes in Urinary Albumin-to-Creatinine Ratio (UACR)
Description: Urinary Albumin-to-Creatinine Ratio from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: Baseline and Week 2, 6, 12, 16 (Follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 43 | 44
mg/g
  Visit 4 (Week 2) | 25.44 (69.166) | 53.88 (68.229) | -86.20 (67.932)
  Visit 5 (Week 6) | -81.90 (68.156) | -30.37 (67.233) | -86.12 (66.940)
  Visit 6/ET (Week 12) | 61.92 (92.291) | -40.10 (91.041) | -135.57 (90.645)
  Visit 7/ Follow up (Week 16) | 72.07 (90.045) | 58.31 (88.825) | -8.27 (88.439)
Statistical Analysis 1: Comparison: TMX-049 Placebo vs TMX-049 40 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3955, ANCOVA; LS Mean Difference = -102.02, 95% CI 2-sided [-338.81 to 134.78]
Statistical Analysis 2: Comparison: TMX-049 Placebo vs TMX-049 200 mg QD; For Week 12 (visit of the primary outcome), ANCOVA model with treatment, randomization strata of UACR levels as independent variables is fitted. The last observation carried forward imputation was used for missing data; Test type: Superiority; p = 0.0991, ANCOVA; LS Mean Difference = -197.49, 95% CI 2-sided [-432.73 to 37.75]

5. Secondary Outcome: Proportion of Subjects With a Greater Than 30% Reduction From Baseline to Week 12 in Urinary Albumin-to-Creatinine Ratio
Description: Changes in Proportion of Subjects With a Greater Than 30% Reduction From Baseline to Week 12 in Urinary Albumin-to-Creatinine Ratio were measured. Subject with greater than 30% reduction is estimated as responder, less than or equal to 30% reduction is estimated as non-responder.
Time Frame: 16 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 43 | 44
Participants
  Responder | 10 | 14 | 19
  Non-responder | 32 | 29 | 25
Statistical Analysis 1: Comparison: TMX-049 Placebo; Odds ratio, 95% CLs, and p-values are obtained from logistic regression model adjusting for treatment group, randomization strata of Baseline sUA (<6.0 vs ≥6.0 mg/dL) and Baseline UACR (200 to <300 mg/g vs 300 to ≤3000 mg/g), Baseline UACR and Baseline sUA levels. Odds ratio for a baseline covariate is the ratio of odds over one unit increase of the covariate and it is assumed constant. P-value represents the statistical significance level of odds ratio differing from 1; Test type: Superiority; p = 0.2791, Regression, Logistic; Odds Ratio (OR) = 1.72 — Missing observations at Study Week 12 are imputed as nonresponse
Statistical Analysis 2: Comparison: TMX-049 Placebo vs TMX-049 200 mg QD; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0507, Regression, Logistic; Odds Ratio (OR) = 2.57

6. Secondary Outcome: Changes in Exploratory Blood Biomarkers (C Reactive Protein)
Description: Changes in Exploratory Blood Biomarkers for inflammation (C Reactive Protein) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: Safety Population consisted of all randomized subjects who received at least one study drug tablet or capsule. Subjects were analyzed according to the actual treatment received.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 42 | 42 | 43
  Visit 4 (Week 2) | 0.046 (0.5168) | 0.014 (0.5384) | 0.087 (0.6194)
  Visit 5 (Week 6): number analyzed (Participants) | 42 | 43 | 42
  Visit 5 (Week 6) | -0.011 (0.6443) | 0.003 (0.3688) | -0.084 (0.4303)
  Visit 6/ET (Week 12): number analyzed (Participants) | 41 | 42 | 42
  Visit 6/ET (Week 12) | 0.000 (0.7527) | -0.144 (0.3691) | 0.000 (0.5176)
  Visit 7/ Follow up (Week 16): number analyzed (Participants) | 41 | 43 | 40
  Visit 7/ Follow up (Week 16) | 0.012 (0.6507) | -0.084 (0.3606) | -0.046 (0.3917)

7. Secondary Outcome: Changes in Exploratory Blood Biomarkers (Soluble TNF Receptor Type I)
Description: Changes in Exploratory Blood Biomarkers for inflammation (Soluble TNF [tumor necrosis factor] Receptor Type I) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- for 12 weeksTMX-049 Placebo: Placebo: Matching placebo to be taken orally, once daily for 12 weeks
Arm/Group | for 12 weeksTMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
ng/L
  Visit 4 (Week 2): number analyzed (Participants) | 42 | 42 | 44
  Visit 4 (Week 2) | -13.7 (367.11) | -92.3 (298.83) | 38.7 (360.03)
  Visit 5 (Week 6): number analyzed (Participants) | 42 | 43 | 43
  Visit 5 (Week 6) | -77.1 (295.50) | 47.6 (485.92) | 60.7 (397.76)
  Visit 6 (Week 12): number analyzed (Participants) | 41 | 42 | 43
  Visit 6 (Week 12) | 16.5 (371.88) | 10.8 (455.11) | 43.8 (265.35)
  Visit 7/Follow up (Week 16): number analyzed (Participants) | 41 | 43 | 42
  Visit 7/Follow up (Week 16) | -25.8 (366.94) | -36.3 (308.79) | 13.8 (320.22)

8. Secondary Outcome: Changes in Exploratory Renal Biomarkers (Creatinine-Corrected Fatty Acid Binding Protein 1)
Description: Changes in Exploratory Renal Biomarkers for renal tubular diseases (Creatinine-Corrected Fatty Acid Binding Protein 1) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L/mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
ug/L/mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 37 | 36 | 33
  Visit 4 (Week 2) | 0.03 (0.161) | 0.01 (0.214) | -0.04 (0.201)
  Visit 5 (Week 6): number analyzed (Participants) | 37 | 37 | 31
  Visit 5 (Week 6) | -0.04 (0.309) | 0.04 (0.258) | -0.04 (0.201)
  Visit 6 (Week 12): number analyzed (Participants) | 37 | 36 | 34
  Visit 6 (Week 12) | -0.01 (0.317) | -0.01 (0.136) | -0.01 (0.218)
  Visit 7/Follow up (Week 16): number analyzed (Participants) | 36 | 36 | 28
  Visit 7/Follow up (Week 16) | 0.02 (0.321) | 0.04 (0.289) | 0.00 (0.188)

9. Secondary Outcome: Changes in Exploratory Renal Biomarkers (Creatinine-Corrected Hydroxy Deoxyguanosine)
Description: Changes in Exploratory Renal Biomarkers for renal tubular diseases (Creatinine-Corrected Hydroxy Deoxyguanosine) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nmol/L/mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
nmol/L/mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 23 | 28 | 31
  Visit 4 (Week 2) | 1.47 (4.266) | 4.70 (4.123) | 6.08 (5.809)
  Visit 5 (Week 6): number analyzed (Participants) | 19 | 25 | 31
  Visit 5 (Week 6) | 1.72 (5.179) | 3.22 (5.321) | 4.88 (5.930)
  Visit 6 (Week 12): number analyzed (Participants) | 18 | 28 | 32
  Visit 6 (Week 12) | -1.86 (5.372) | 3.75 (6.157) | 6.87 (10.476)
  Visit 7/ Follow up (Week 16): number analyzed (Participants) | 19 | 27 | 23
  Visit 7/ Follow up (Week 16) | 1.20 (5.480) | -0.07 (5.647) | -3.14 (5.211)

10. Secondary Outcome: Changes in Exploratory Renal Biomarkers (Creatinine-Corrected Kidney Injury Molecule-1)
Description: Changes in Exploratory Renal Biomarkers for renal tubular diseases (Creatinine-Corrected Kidney Injury Molecule-1) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L/mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
ug/L/mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 40 | 39 | 41
  Visit 4 (Week 2) | 0.00 (0.010) | 0.00 (0.016) | 0.00 (0.007)
  Visit 5 (Week 6): number analyzed (Participants) | 38 | 39 | 39
  Visit 5 (Week 6) | 0.00 (0.010) | 0.00 (0.015) | 0.00 (0.006)
  Visit 6 (Week 12): number analyzed (Participants) | 39 | 40 | 41
  Visit 6 (Week 12) | 0.00 (0.019) | 0.00 (0.015) | 0.00 (0.008)
  Visit 7/Follow up (Week 16): number analyzed (Participants) | 39 | 40 | 38
  Visit 7/Follow up (Week 16) | 0.00 (0.009) | 0.00 (0.0014) | 0.00 (0.009)

11. Secondary Outcome: Changes in Exploratory Renal Biomarkers (Creatinine-Corrected N-acetyl-beta-D-glucosaminidase)
Description: Changes in Exploratory Renal Biomarkers for renal tubular diseases (Creatinine-Corrected N-acetyl-beta-D-glucosaminidase) from Baseline to Weeks 2, 6, 12/early termination, and 16 (Follow-up) were measured.
Time Frame: 16 Weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L/mg/dL
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049 200 mg QD
Number analyzed (Participants) | 42 | 44 | 44
U/L/mg/dL
  Visit 4 (Week 2): number analyzed (Participants) | 41 | 43 | 44
  Visit 4 (Week 2) | -0.01 (0.129) | 0.03 (0.136) | -0.01 (0.152)
  Visit 5 (Week 6): number analyzed (Participants) | 41 | 42 | 41
  Visit 5 (Week 6) | 0.02 (0.154) | 0.02 (0.121) | -0.02 (0.147)
  Visit 6 (Week 12): number analyzed (Participants) | 40 | 41 | 43
  Visit 6 (Week 12) | 0.00 (0.123) | 0.02 (0.143) | -0.02 (0.108)
  Visit 7/Follow up (Week 16): number analyzed (Participants) | 39 | 42 | 40
  Visit 7/Follow up (Week 16) | 0.01 (0.089) | 0.02 (0.116) | -0.01 (0.132)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) reporting began from the time of informed consent and ends at the Follow-up Visit (Visit 7), up to 16 weeks. For subjects without the Follow-up Visit, the reporting ends 28 days after the last dose of the Investigational Medicinal Product, up to 12 weeks.
Description: Treatment-emergent AEs (TEAEs) were defined as any events with start date on or after the date of first dose of double-blind study drug and up to 30 days after date of last dose of double-blind study drug.
Groups:
- TMX-049: 200 mg: TMX-049: 200 mg of TMX-049 to be taken orally, once daily
Arm/Group | TMX-049 Placebo | TMX-049 40 mg QD | TMX-049: 200 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 4/42 | 4/44 | 2/44
Other Adverse Events (participants affected / at risk) | 18/42 | 19/44 | 17/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMX-049 Placebo (N=42) | TMX-049 40 mg QD (N=44) | TMX-049: 200 mg (N=44)
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMX-049 Placebo (N=42) | TMX-049 40 mg QD (N=44) | TMX-049: 200 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Reticulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0
Middle ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 3
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0
Drug interaction (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 2 | 0
Oedema peripheral (General disorders) | 1 | 3 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 2
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Haematology test abnormal (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03449199/Prot_002.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03449199/SAP_003.pdf